CLINICAL TRIAL: NCT03846791
Title: An Evaluation of Health Outcomes for Mako Hip Replacement
Acronym: HELLO
Status: Completed | Type: Observational
Sponsor: Bournemouth University (Other)
Collaborators: Nuffield Health Bournemouth (Unknown); Orthopaedic Research Institute (Unknown); Stryker Orthopaedics (Industry)
Responsible Party: Sponsor
Other Study IDs: ORI/Mako/18
Record Dates: First submitted 2019-02-13; First posted 2019-02-20 (Actual); Last update posted 2024-08-13 (Actual); Status verified 2024-08

CONDITIONS: Osteoarthritis, Hip
MeSH Terms: conditions — Osteoarthritis, Hip

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Observational Study Post MAKO Robotic Surgery — To assess clinical outcomes and surgery related resource use in the year post surgery for patients undergoing hip replacement surgery using the MAKO robot

SUMMARY:
To assess clinical outcomes and surgery related resource use in the year post surgery for patients undergoing hip replacement using the Mako Robo

DETAILED DESCRIPTION:
This is an observational cohort study. It evaluates the recovery of 200 patients who are having routine robotic hip replacement surgery at a Nuffield Hospital in Bournemouth. Any complications from the surgery, or readmissions to hospital, will be reported. Investigators will measure how accurately the surgeon, assisted by the robotic-arm, positions the hip implant during the surgery using x-rays taken as part of routine care. The study also monitors the progress of rehabilitation by assessing pain and functional ability in the year following surgery, and will investigate whether there is an association between this recovery and a measurement of an area of muscle in the pelvic region, taken from a routine CT scan.

Patients will be asked to come to the Orthopaedic Research Institute at Bournemouth University to be assessed before they have surgery, and again at 3 weeks, 6-8 weeks, 3 months, 6 months and 12 months following surgery. At these visits they will be asked about their pain, how well they can do daily activities, and their quality of life. They will be assessed on their ability to sit-to-stand five times, walk for 40m, and climb some stairs. At each visit, except the three weeks visit, they will also have their gait tested on a specialised clinical treadmill, and the muscle strength in their legs measured. They will also be measured for oedema at baseline, 3 weeks and 6-8 weeks using a Fit3D ProScanner. These visits are in addition to the routine clinical follow-up visits at Nuffield Hospital. Participants will also be invited to wear a wrist activity monitor for at least three consecutive days prior to surgery and for the 6 weeks following discharge so that their activity can be recorded.

Surgery-related resource use of the procedure will also be reported, such as length of hospital stay, time in theatre, unplanned hospital visits, non-routine medication, outpatient appointments and physiotherapy appointments.

ELIGIBILITY:
Inclusion Criteria:

* Non-inflammatory degenerative joint disease including osteoarthritis and avascular necrosis, suitable for unilateral primary hip replacement;
* Rheumatoid arthritis;
* Correction of functional deformity;
* Voluntary written Informed Consent obtained.
* Participant able to complete study follow-up.

Exclusion Criteria:

* Prospect for recovery to independent mobility compromised by known coexistent medical problems;
* Requiring revision hip replacement;
* Previous hip replacement (resurfacing or THR) on the contralateral side, with outcome achieving an Oxford Hip score <18 points;
* Likely post-operative leg length inequality >5cm;
* Neuromuscular disease affecting hip (Parkinson's, cerebral palsy, other spasticity);
* Primary or metastatic tumor involving this hip;
* Loss of abductor musculature, poor bone stock, or poor skin coverage around the hip joint;
* Previous arthrodesis or excision arthroplasty
* Acetabular deficiency - >2cm superior loss acetabular dome or >1.5cm protrusion acetabulae or wall deficiency> half a wall;
* Dysplasia (DDH) with >2.5cm subluxation or complete dislocation;
* Body mass index > 40kg/m2;
* Active or previous or suspected infection in this hip;
* Sepsis or osteomyelitis;
* Known sensitivity to device materials;
* Not physically able to use Grail gait lab and Primus muscle testing equipment;
* Women judged by the Investigator to be of childbearing potential who are pregnant, nursing, or planning to become pregnant, and those who do not agree to remain on an acceptable method of birth control throughout the entire study period;
* Unable to provide informed consent (insufficient English, cognitive disorder such as dementia, psychiatric illness);
* Unable to complete follow-ups (life expectancy <5 years, insufficient English, lives overseas, unable to return easily).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing Robot Assisted Total Hip Replacement at the Nuffield Health
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2019-07-15 (Actual); Primary Completion 2024-05-03 (Actual); Study Completion 2024-05-03 (Actual)

PRIMARY OUTCOMES:
The measurement of surgical complications post surgery | 1 Year post surgery
  This study's primary outcome is to report on surgical complications. Events will be sub-classified as device (prosthesis or robot) or surgeon related.
The measurement of readmission post surgery | 1 Year post surgery
  This study's primary outcome is to report on surgical complications. Events will be sub-classified as device (prosthesis or robot) or surgeon related.

SECONDARY OUTCOMES:
Accuracy of component positioning | 1 Year post surgery
  Placement of prosthetic components will be evaluated by assessing radiographs
Functional Assessments - Chair stand | 1 Year post surgery
  30 s Chair Stand test as recommended by the Osteoarthritis Research Society International (OARSI). Assessment will be done prior to surgery, and again at 3 weeks, 6-8 weeks, 3 months, 6 months and 1 year following surgery
Functional Assessments - Fast paced Walk | 1 Year post surgery
  40m fast-paced walk test as recommended by the Osteoarthritis Research Society International (OARSI). Assessment will be done prior to surgery, and again at 3 weeks, 6-8 weeks, 3 months, 6 months and 1 year following surgery
Functional Assessments - Stair Climb | 1 Year post surgery
  Stair climb test as recommended by the Osteoarthritis Research Society International (OARSI). Assessment will be done prior to surgery, and again at 3 weeks, 6-8 weeks, 3 months, 6 months and 1 year following surgery
Gait analysis | 1 Year post surgery
  Participants' gait will be analysed using the GRAIL MotekForce at baseline, 6-8 weeks, 3 months, 6 months and 1 year following surgery.
Muscle Testing | 1 Year post surgery
  Participants' muscle strength will be analysed using the Primus BTE at baseline, 6-8 weeks, 3 months, 6 months and 1 year following surgery.
Measurement of pre-operative psoas muscle mass | Pre-Operative
  This measurement will be taken from the pre-surgery CT scan
Patient Reported Outcome Measures - EQ-5D Quality of Life Score | 6 Months post surgery
  EQ-5D Quality of Life Score will be assessed at pre-surgery and at 6 months.
Patient Reported Outcome Measures - The Pain Catastrophizing Score (PCS) | Pre-Operative
  The Pain Catastrophizing Score (PCS) will be assessed prior to surgery.
Patient Reported Outcome Measures - The Hip Disability and Osteoarthritis Outcome Score (HOOS) | 1 Year post surgery
  The Hip Disability and Osteoarthritis Outcome Score (HOOS) will be assessed at pre-surgery, 3 weeks, 6-8 weeks, 3 month, 6 months and 1 year following surgery
Surgery related resource use - length of stay in hospital | 1 Year post surgery
  Data will be reported on surgery-related use of resources for length of stay in hospital
Surgery related resource use - time in theatre | 1 Year post surgery
  Data will be reported on surgery-related use of resources for time in theatre
Surgery related resource use - unplanned hospital visits | 1 Year post surgery
  Data will be reported on surgery-related use of resources for unplanned hospital visits
Surgery related resource use - non-routine medication | 1 Year post surgery
  Data will be reported on surgery-related use of resources for non-routine medication
Surgery related resource use - number of outpatient appointments | 1 Year post surgery
  Data will be reported on surgery-related use of resources for number of outpatient appointments
Surgery related resource use - number of physiotherapy appointments | 1 Year post surgery
  Data will be reported on surgery-related use of resources for number of physiotherapy appointments.
Monitoring of physical activity | 6-8 weeks following surgery
  Participants will be invited to wear an activity monitor on their wrist for at least three consecutive days prior to surgery, and for the 6-8 weeks following discharge
Measurement of oedema | 6-8 weeks following surgery
  Participants will be assessed for oedema using a Fit3D ProScanner at baseline, 3 weeks and 6-8 weeks following surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Tom Wainwright, Study Director — Professor
Locations (2):
- United Kingdom (2):
  - Nuffield Health Bournemouth, Bournemouth
  - Orthopaedic Research Institute Bournemouth University, Bournemouth

IPD SHARING:
Plan to Share IPD: No